CLINICAL TRIAL: NCT02211027
Title: Active Immunization of Patients With Head and Neck Squamous Cell Carcinoma (HNSCC) Using Fibroblasts Transfected With DNA From Autologous Tumor
Brief Title: Biological Vaccine: Semi-allogeneic Human Fibroblasts (MRC-5) Transfected With DNA
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Robert Ferris (Other)
Collaborators: Immune Cell Therapy Inc. (Industry)
Responsible Party: Sponsor-Investigator, Robert Ferris, Professor of Otolaryngology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-160
Record Dates: First submitted 2014-07-16; First posted 2014-08-07 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Head and Neck Squamous Cell Carcinoma (HNSCC)
Keywords: Squamous Cell Carcinoma; Head & Neck Cancer; Vaccine; Carcinoma; Immunization; Autologous Tumor
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell; Head and Neck Neoplasms; Carcinoma | interventions — DNA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaccine (Experimental): The vaccine is composed of lethally irradiated semi-allogenic human fibroblasts (MRC-5) transfected with genomic tumor DNA from the patients own tumor.
  Interventions: Biological: Semi-allogenic human fibroblast (MRC-5) transfected with DNA

INTERVENTIONS:
Biological: Semi-allogenic human fibroblast (MRC-5) transfected with DNA — Each vaccination consists of up to 1 x 10e7 (not less than 7 x 10e6) DNA-transfected irradiated fibroblasts. Each vaccination will be administered intradermally using a 1 mL syringe and a 25 gauge needle.The first immunization will be administered at least 12 weeks after surgery or completion of adjuvant chemotherapy and/or radiotherapy.Three additional vaccines will be administered once a week for a total of four vaccines.
  Patients will have vaccinations administered at 4 different sites as follows:
  Site #1: Right arm Site #2: Left arm Site #3: Right thigh Site #4: Left thigh. Approximately equal numbers of transfected fibroblasts will be administered at each site.

SUMMARY:
Hypothesis The incidence of toxicity in patients receiving the tumor DNA-transfected fibroblast vaccine will be acceptably low and the immunologic response rate sufficiently high to warrant further study of this therapy

The study of the vaccine will proceed in two stages after the method of Simon (102). In the first stage, 15 patients will be accrued and treated. If two or fewer objective immunologic responses occur, the study will be terminated. If 3 or more responses are observed, the study will proceed to the second stage, accruing an additional 22 patients. If the second stage is complete and a total of 9 or more immunologic responses are observed among the 37 patients treated, the treatment response rate for the vaccine will be considered high enough to warrant further study. Conversely, if the evaluation of the vaccine concludes at the first stage, or if 8 or fewer total immunologic responses occur after completing the second stage, the vaccine will not be considered for further study.

DETAILED DESCRIPTION:
This is a single institution open-label phase Ib clinical trial designed to determine the safety of immunization of patients with resected Head and Neck Squamous Cell Carcinoma (HNSCC) with lethally irradiated semi-allogeneic human fibroblasts (MRC-5) transfected with DNA derived from the subject's own tumor and to measure the immune response to the autologous tumor vaccine.

Briefly, the plan is to use a two-stage trial design and to initially enroll 15 patients with Head and Neck Squamous Cell Carcinoma (HNSCC). The patients will undergo surgical resection to provide complete removal of the primary lesion with negative gross and microscopic margins. A portion of the primary tumor specimen not necessary for the pathologic diagnosis will be obtained to serve as a source of DNA for preparing the vaccine. Each DNA-based vaccine will contain 1 x 10e7 DNA-transfected human allogeneic fibroblasts. The vaccine will be lethally irradiated before it is used for immunization. It will be administered intradermally in the Outpatient Clinic for a total of four vaccinations delivered at weekly intervals.

Patients delayed-type hypersensitivity (DTH) responses will be tested but will not be an eligibility criterion. Immunologic response to the vaccine will be evaluated. If there is no evidence of toxicity, and >3 of the 15 initial patients show immunologic response, the second stage of the study will be opened for accrual of 22 patients.

To determine patient's response to the DNA-based vaccines, the frequency of T cells reactive with recipient cells transfected with the autologous tumor DNA will be measured by ELISPOT for IFN-y and compared with the response to non-transfected fibroblasts prior to and after vaccination. All patients will be monitored for Immunologic response by assays include ELISPOT, flow cytometry for lymphocyte markers, Annexin V binding, TcR expression, caspase3 activity and serum antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Pathological stage I-IVa HNSCC
* The subject must have a complete removal of the primary HNSCC lesion with negative gross and microscopic margins. Documentation of margins by frozen sections at surgery is recommended. Patients who have already had surgery and have available banked tumor samples can be enrolled AFTER surgery.
* At least 18 years of age.
* Karnofsky performance status >/= 70
* Adequate hematologic function:
* Absolute neutrophil count > 1,000/mm3
* Absolute lymphocyte count > 1,000/mm3
* Hemoglobin > 9 g/dL
* Platelets > 100,000/mm3
* Liver function tests:
* Bilirubin (total) < /=1.7 mg/dL
* Alkaline phosphatase < 252 u/L
* SGOT < 108 u/L
* Kidney profile:
* Serum electrolytes
* Sodium 136-146 mEq/L
* Potassium 3.5-5.0 mEq/L
* Bicarbonate 21-31 mEq/L
* Chloride 98-107 mmol/L
* Serum creatinine < 3 x ULN
* BUN 8-26 mg/dL
* At least a 12 week interval should have elapsed between prior surgery, radiation therapy, chemotherapy or any other treatment and the first vaccination. Patients should have recovered from surgery and adjuvant treatment.
* The effects of the tumor DNA-transfected fibroblast vaccine on the developing human fetus are unknown. For this reason women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for 4 months after the last dose of the study vaccine, even if oral contraceptives are used. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of the tumor DNA-transfected fibroblast vaccine administration.

Exclusion Criteria:

Patients will be EXCLUDED from participation in the study if any of the following apply:

* One or more of the Inclusion Criteria are not met.
* A significant history or current evidence of cardiac disease including, but not limited to: congestive heart failure, coronary artery disease, angina pectoris, uncontrolled hypertension, serious arrhythmias or myocardial infarction within the previous six months.
* Evidence of ongoing or active infection requiring antibiotic therapy.
* Active intracranial metastases. Patients with previously resected intracranial disease and/or previously irradiated intracranial metastases that have been clinically stable for four weeks are eligible.
* Pregnant or lactating women. Pregnant women are excluded from this study. Women of childbearing potential must have a negative pregnancy test per standard of care prior to the surgery for tumor removal. A second pregnancy test must be performed 7 days prior to the first vaccination and must be negative. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued if the mother is treated on study.
* Patients requiring systemic corticosteroids (unless patients have had no corticosteroids within 4 weeks prior to start of study).
* Autoimmune disease including, but not limited to, rheumatoid arthritis, systemic lupus erythematous, multiple sclerosis, or ankylosing spondylitis.
* Patients who have post-obstructive pneumonia or other serious infection at the time of registration or other serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the patient has been disease-free for at least 5 years prior to registration.
* Uncontrolled intercurrent illness including, but not limited to psychiatric illness/social situations that would limit compliance with study requirements.
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study. HIV testing will be performed in patients receiving combination anti-retroviral therapy when indicated per medical records review.
* Patients with clinical symptoms of Hepatitis B and/or Hepatitis C will be tested, if clinically indicated per medical records review. Positive results will be an exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2017-10 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Immunization Safety | 2.5 years
  Toxicity will be monitored continuously from the first vaccination through the 6 month post follow up study visit for each subject.
  Patients will have a follow-up visit at 1 week after last vaccination (day 29, off treatment), at 1 month, 3 months and 6 months after last vaccination or after removal from study or until death, whichever occurs first. After the 6 month follow-up visit, subjects will be followed for survival only (no additional clinical trial site visits). Patients removed from study for unacceptable adverse event(s) will be followed until resolution or stabilization of the adverse event.
  All subjects should be enrolled within 2 years and follow up studies complete within 3 years.

SECONDARY OUTCOMES:
Immunologic Response Rate to the the tumor DNA-transfected fibroblast vaccine | 2.5 years
  Immunologic evidence of a response to the DNA-based vaccine will depend on the results of ELISPOT assays performed at five to seven time points: pre-surgery, pre-vaccine (either at the day -28 or Day 1 prior to vaccination), on day 15, on day 29, 1 month, 3 months (if clinically indicated at 1 and 3 months) and at the 6 month post treatment follow-up appointment. A significant difference in the frequency of vaccine reactive or anti-tumor-reactive T cells between pre- and post-vaccine determinations will be considered as a positive immune response to the vaccine.
  Additionally, immune competence and the presence/absence of immune suppression will be evaluated before and after vaccine administration. The ability of DNA-based vaccines to reverse or diminish demonstrated effects in signaling defects, lymphocyte apoptosis or proportions of T(reg) in the peripheral circulation will be measured but will not be used as a criterion for evaluation of the immune response.

OTHER OUTCOMES:
Immune competence | 2.5 years
  Immune competence and the presence/absence of immune suppression will be evaluated before and after vaccine administration and at the 6 month follow-up visit. The ability of DNA-based vaccines to reverse or diminish demonstrated effects in signaling defects, lymphocyte apoptosis or proportions of T(reg) in the peripheral circulation will be measured but will not be used as a criterion for evaluation of the immune response.

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Ferris, MD, Principal Investigator — Professor of Otolaryngology, Eye & Ear Institute of the University of Pittsburgh Medical Center.
Locations (3):
- United States (3):
  - University of Pittsburgh Medical Center Presbyterian Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute-Hillman Cancer Center, Pittsburgh, Pennsylvania
  - University Of Pittsburgh Medical Center- Shadyside Hospital, Pittsburgh, Pennsylvania